CLINICAL TRIAL: NCT05956028
Title: Efficacy of Ultrasound-guided Internal Jugular Vein Versus Supraclavicular Subclavian Vein Cannulation in Neonates and Infants Less Than 5 kg Undergoing Major Surgeries: a Prospective, Randomized Controlled Trial.
Brief Title: Efficacy of Ultrasound-guided Internal Jugular Vein Versus Supraclavicular Subclavian Vein Cannulation in Neonates and Infants Less Than 5 kg.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kasr El Aini Hospital (Other)
Responsible Party: Principal Investigator, Khaled Abdelfattah Abdallah Sarhan, principal investigator, Asst. professor of anesthesia, Cairo university, Kasr El Aini Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MD-159-2023
Record Dates: First submitted 2023-07-13; First posted 2023-07-21 (Actual); Last update posted 2025-03-04 (Actual); Status verified 2025-03

CONDITIONS: Pediatric; Anesthesia; Central Venous Catheter; Ultrasound; Internal Jugular Vein
Keywords: ultrasound; central venous catheter; neonates; subclavian vein; internal jugular vein; anesthesia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- (group S) (Experimental): receive ultrasound guided subclavian vein cannulation
  Interventions: Procedure: Ultrasound guided SCV cannulation; Procedure: Ultrasound guided IJV cannulation
- (group I) (Active Comparator): receive ultrasound guided internal jugular vein cannulation
  Interventions: Procedure: Ultrasound guided SCV cannulation; Procedure: Ultrasound guided IJV cannulation

INTERVENTIONS:
Procedure: Ultrasound guided SCV cannulation — receive ultrasound guided SCV cannulation
Procedure: Ultrasound guided IJV cannulation — receive ultrasound guided IJV cannulation

SUMMARY:
The aim of this study is to compare the effectiveness and safety of ultrasound- guided IJV and supraclavicular SCV cannulation in infants weighing less than 5 kg.

DETAILED DESCRIPTION:
The aim of this study is to compare the effectiveness and safety of ultrasound- guided IJV and supraclavicular SCV cannulation in infants weighing less than 5 kg.

It is hypothesized that ultrasound guided supraclavicular SCV cannulation has a higher success rate compared to IJV cannulation.

Infants will be recruited into the trial during pre-operative assessment. Recruited infants will be randomly assigned to one of two groups in a 1:1 ratio; (group S) to receive ultrasound guided SCV cannulation and (group I) to receive ultrasound guided IJV cannulation. Randomization will be achieved using a computer-generated sequence. Concealment will be achieved using opaque envelopes.

All infants will be anesthetized in accordance with the local policy of pediatric anesthesia unit in Abu El-Reesh pediatric hospital-Cairo university after ethics committee approval.

After preoperative examination and upon arrival to the operating room heart rate, noninvasive blood pressure NBP and oxygen saturation SPO2 will be monitored using standard monitor (drȁger infinity vista XL) before inhalational induction of anesthesia using titration of sevoflurane in oxygen air mixture 60% (starting from 3% up to 8%) until the infant is put to sleep. After securing an intravenous line anesthesia will be completed with 1-2µg/kg of fentanyl and atracurium 0.5 mg/kg.

Induction of anesthesia will be performed by the attending senior anesthesia resident who has finished at least 2 years of residency (who is independent of the study team).

All cannulations will be performed by 2 pediatric anesthesiologists trained in US-guided central line placement each one has performed (more than 50 cannulations) before the study. Catheterization will be performed using a standard Seldinger technique under sterile conditions using high frequency (5-10 MHz) footprint ultrasound probe (S-NerveTM; SonoSite Inc., Bothell, WA, USA).

Before the procedure, IJV or SCV veins size, patency, and collapsibility with transducer pressure will be assessed using US probe. The cannulation side (right or left) choice and the central venous catheter size will be decided by the practitioner preference according to the patient's vein examination.

Group I:

The standard transverse out-of-plane approach will be used. Infants will be placed in the 10° Trendelenburg and a shoulder roll will be placed to extend the neck, which will be rotated about 30° to the opposite side of cannulation. The transducer will be placed in a transverse position over the patient's neck at the level of cricoid cartilage to identify IJV and common carotid artery (CCA) in short-axis view. The CCA and the IJV will be differentiated by pulsations of the artery and compressibility of the vein. The vein will be then centered on the screen. The skin puncture will be made in the center of the US image using a needle without syringe. The needle will be introduced at an angle of 60° to the skin surface, perpendicular to the transducer. The needle will be advanced toward IJV until an indentation of the anterior wall of the vein is noticed. If spontaneous blood flashback is obtained, the guide wire will be introduced into the vein and the procedure will be completed using Seldinger's technique. If no spontaneous blood return is observed despite clear visualization of the needle bevel in the vessel lumen on US, a syringe will be attached to the needle hub to aspirate blood and then the guide wire will be introduced into the vein and the procedure will be completed. The attempt will be considered successful when smooth insertion of the guidewire into the vein after confirmation of the site of the wire in the right atrium using intraoperative x ray. If blood could not be aspirated, the needle will be withdrawn, the attempt will be considered failed and another attempt will be made to a maximum of 3 attempts. If failure more than 3 attempts, another site will be chosen and the patient will be excluded from the study.

Group S:

The patient will be positioned with the neck extended and rotated 45° opposite to the cannulation side. A towel roll will be placed under the shoulders for adequate neck extension. The US probe will be placed against and above the clavicle to visualize the transversal view of carotid artery and IJV, and then will be slowly tilted against the infant's cheek, showing first the subclavian artery in longitudinal view, and then, more anterior, the SCV, lying on the pleural line.

After obtaining a satisfactory image of the SCV in the longitudinal axis, the needle will be introduced without syringe in an in-plane technique. If spontaneous blood flashback is obtained, the guide wire will be introduced into the vein and the procedure will be completed using Seldinger's technique. If no spontaneous blood return is observed despite clear visualization of the needle bevel in the vessel lumen on US, a syringe will be attached to the needle hub to aspirate blood and then the guide wire will be introduced into the vein and the procedure will be completed. The attempt will be considered successful when smooth insertion of the guidewire into the vein after confirmation of the site of the wire in the right atrium using intraoperative x ray. If blood could not be aspirated, the needle will be withdrawn, the attempt will be considered failed and another attempt will be made. If failure more than 3 attempts, another site will be chosen, and the patient will be excluded from the study.

ELIGIBILITY:
Inclusion Criteria:

* • All infants weighing less than 5 kg scheduled for major elective surgeries under general anesthesia.

Exclusion Criteria:

* • Parents or legally authorized personnel refusal.

  * Previous trials of central venous cannulation in the last week.
  * Emergency surgery.
  * Coagulopathy (platelets less than 20.000 and or INR more than 1.5)
  * Infection at the proposed site for cannulation.
  * Inability to visualize vein correctly by the ultrasound.
  * Neck deformity or swelling in the proposed site of cannulation.

Ages: 1 Day to 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 108 (Actual)
Dates: Start 2023-07-21 (Actual); Primary Completion 2025-03-03 (Actual); Study Completion 2025-03-03 (Actual)

PRIMARY OUTCOMES:
The first attempt success rate. | 1 hour
  The attempt will be considered successful when smooth insertion of the guidewire into the vein.

SECONDARY OUTCOMES:
Insertion time | 1 hour
  defined as time from the start of the needle puncture till smooth insertion of the guide wire
Number of puncture attempts. | 1 hour
  Number of puncture attempts.

CONTACTS AND LOCATIONS:
Overall Officials: Khaled Sarhan, Principal Investigator — Cairo University
Locations (1):
- Cairo university hospitals, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sarhan K, Abdelgawad O, Abdelhamid B, El-Ashmawi H, Soliman D, Turki D, Salah H, Badry M. Efficacy of Ultrasound-Guided Internal Jugular Vein versus Subclavian Vein Cannulation in Neonates and Infants Weighing Less Than 5 kg: A Prospective, Randomized Controlled Trial. Anaesth Crit Care Pain Med. 2025 Nov 17:101681. doi: 10.1016/j.accpm.2025.101681. Online ahead of print. PMID 41260395